CLINICAL TRIAL: NCT00867997
Title: Noncarious Cervical Lesion Treatment Outcomes: Randomized Clinical Trial
Brief Title: Noncarious Cervical Lesion Treatment Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRL0707; U01DE016755 (NIH); 116358
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Noncarious Cervical Lesions
Keywords: Noncarious Cervical Lesions; Hypersensitivity; Teeth; Dentistry; Practice-based research network
MeSH Terms: conditions — Hypersensitivity | interventions — Clearfil S3 Bond

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dentifrice (Active Comparator): Chemoactive (remineralizing, neuroactive) dentifrice treatment
  Interventions: Other: Chemoactive (remineralizing, neuroactive) dentifrice treatment
- Sealant (Active Comparator): DBA/sealant application
  Interventions: Other: Clearfil S3 Bond; Clearfil Liner Bond 2 Protect Liner F
- Resin-based composite (Active Comparator): Restoration with a dentin bonding agent (DBA) and flowable resin-based composite
  Interventions: Other: Clearfil S3 Bond; Premise Flowable resin-based composite

INTERVENTIONS:
Other: Chemoactive (remineralizing, neuroactive) dentifrice treatment — Chemoactive (remineralizing, neuroactive) dentifrice treatment
  Arms: Dentifrice
Other: Clearfil S3 Bond; Clearfil Liner Bond 2 Protect Liner F — Self-etch DBA followed by a hydrophobic resin layer
  Arms: Sealant
Other: Clearfil S3 Bond; Premise Flowable resin-based composite — Restoration with a dentin bonding agent (DBA) and flowable resin-based composite
  Arms: Resin-based composite

SUMMARY:
The overall objective of this three-armed randomized clinical trial (RCT) is to determine the comparative efficacy of three treatments for hypersensitive noncarious cervical lesions (NCLs): chemoactive dentifrice use, dentin bonding agent (DBA) with sealing, and flowable resin-based composite restoration. The primary outcomes of this study are the reduction/elimination of hypersensitivity and the effect of treatment as measured by patient-reported outcomes. Secondary outcomes, as determined by laboratory evaluation of intraoral replicas of pre- and posttreatment NCL surfaces, are tubule occlusion, retention of resin coating, retention of restoration, and change in lesion size. Outcomes will be ascertained via the following specific aims:

Specific Aim 1: To compare the reduction of hypersensitivity of study teeth by both measurement and by patient-reported outcomes among three treatment groups.

Specific Aim 2: To recruit subjects with teeth with hypersensitive NCLs, measure baseline sensitivity and subject quality of life, administer one of three different treatments to each of three randomized groups of subjects, and determine immediate posttreatment hypersensitivity.

Specific Aim 3: To compare the degree of tubule occlusion before and after the three treatments and to associate these findings with posttreatment hypersensitivity, patient-reported outcomes, and restoration retention.

Treatment of NCLs remains controversial. Few studies have compared treatment methods or their financial implications. This RCT will determine the reduction of NCL hypersensitivity and patient-reported outcomes over a 6-month period for each of three different treatments. This will be the first practice-based research network RCT to combine objective clinical assessment of NCL treatment patient-reported outcomes with laboratory examination of dentin tubule occlusion and lesion size.

ELIGIBILITY:
Inclusion Criteria:

* A premolar or first molar with an NCL and hypersensitivity of ≥3 as indicated by the subject on the Numeric Pain Assessment Scale (2008 NCCN) with standardized air blast stimulation with no other tooth exhibiting hypersensitivity (≥2 as indicated by the subject on the NPAS) in the same quadrant. If the patient has a tooth in more than one quadrant that meet these criteria then the quadrant selected will be that containing the tooth with the highest hypersensitivity reading. If the sensitivities are the same the quadrant with the lesion with the greatest depth would be selected. If the sensitivities and depth are the same the quadrant with the most convenient restorative access will be selected.
* Teeth with NCL depth of at least 1 mm as measured by placing a periodontal probe (e.g.) into the deepest part of the cervical lesion
* Teeth free of mesial, distal, or buccal restorations (to avoid confounding hypersensitivity)
* Teeth with mobility of <1 mm when manipulated between blunt instruments
* Subject able to follow the study protocol and willing to return for all evaluation appointments
* Subject able to comprehend and sign the written consent form
* Subject 18 years of age or older

Exclusion Criteria:

* Subject who has a medical condition that could interfere with reliable pain reporting
* Subject who is taking a medication that could interfere with reliable pain reporting
* Subject who has taken an analgesic medication (narcotic, NSAID, acetaminophen, salicylic acid) within 24 hr pretreatment
* Subject who is undergoing active orthodontic treatment
* Subject with any of the following: a) Hypersensitive teeth with carious lesions; b) Hypersensitive teeth with buccal vertical cracks in enamel; c) Hypersensitive teeth with an irreversible pulpitis (pain lasting more than 5 sec after stimulation); d) Hypersensitive teeth with full crowns; e) Hypersensitive teeth with partial denture clasps on the facial surface; f) Evidence of inflamed gingival tissue and bleeding on probing in the sextant being considered for treatment as part of the study (the etiology of these lesion is closely related to excessive or improper brushing perhaps with an abrasive dentifrice and there is almost never accumulated plaque associated with the NCL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To compare the reduction of hypersensitivity of study teeth by both measurement and by patient-reported outcomes among three treatment groups. | Baseline, 1, 3 and 6 months

SECONDARY OUTCOMES:
To compare the degree of tubule occlusion before and after the three treatments and to associate these findings with posttreatment hypersensitivity, patient-reported outcomes, and restoration retention. | Baseline, 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Curro, DMD, PhD, Principal Investigator — NYU Langone Health
Locations (17):
- United States (17):
  - Maryann Lehmann, DDS, Darien, Connecticut
  - Ahmad Soolari, D.M.D., Potomac, Maryland
  - Oral Health Center, Southborough, Massachusetts
  - Scott B Schaffer, DMD, Clark, New Jersey
  - Gentle Dental Care, LLC, Edison, New Jersey
  - Dr. Howard Spielman, Plainsboro, New Jersey
  - Drs. Martin & Ferraiolo, Totowa, New Jersey
  - Cynthia Jetter, DMD, Voorhees Township, New Jersey
  - Bay Dental PC, Brooklyn, New York
  - Ying Wong, DDS, New York, New York
  - Martin Man, DMD, New York, New York
  - Kay T. Oen, DDS, Port Chester, New York
  - Janice K. Pliszczak, DDS, Syracuse, New York
  - Susan D. Bernstein, DDS, Cincinnati, Ohio
  - Dr. Jeannette Abboud-Niemczyk, Drexel Hill, Pennsylvania
  - Allan J Horowitz, DMD, King of Prussia, Pennsylvania
  - Dr. Julie Ann Barna, Lewisburg, Pennsylvania

REFERENCES:
- [Background] AASM (2001). The international classification of sleep disorders, revised: diagnosis and coding manual. Westchester, IL: American Academy of Sleep Medicine.
- [Background] Absi EG, Addy M, Adams D. Dentine hypersensitivity. The development and evaluation of a replica technique to study sensitive and non-sensitive cervical dentine. J Clin Periodontol. 1989 Mar;16(3):190-5. doi: 10.1111/j.1600-051x.1989.tb01639.x. PMID 2656768
- [Background] Bader JD, Levitch LC, Shugars DA, Heymann HO, McClure F. How dentists classified and treated non-carious cervical lesions. J Am Dent Assoc. 1993 May;124(5):46-54. doi: 10.14219/jada.archive.1993.0112. PMID 8482781
- [Background] Bader JD, McClure F, Scurria MS, Shugars DA, Heymann HO. Case-control study of non-carious cervical lesions. Community Dent Oral Epidemiol. 1996 Aug;24(4):286-91. doi: 10.1111/j.1600-0528.1996.tb00861.x. PMID 8871039
- [Background] Bartlett DW, Shah P. A critical review of non-carious cervical (wear) lesions and the role of abfraction, erosion, and abrasion. J Dent Res. 2006 Apr;85(4):306-12. doi: 10.1177/154405910608500405. PMID 16567549
- [Background] Burke FJ, Whitehead SA, McCaughey AD. Contemporary concepts in the pathogenesis of the Class V non-carious lesion. Dent Update. 1995 Jan-Feb;22(1):28-32. PMID 7664969
- [Background] Ceruti P, Menicucci G, Mariani GD, Pittoni D, Gassino G. Non carious cervical lesions. A review. Minerva Stomatol. 2006 Jan-Feb;55(1-2):43-57. English, Italian. PMID 16495872
- [Background] Duran I, Sengun A. The long-term effectiveness of five current desensitizing products on cervical dentine sensitivity. J Oral Rehabil. 2004 Apr;31(4):351-6. doi: 10.1046/j.1365-2842.2003.01241.x. PMID 15089941
- [Background] Gillam DG, Newman HN, Davies EH, Bulman JS, Troullos ES, Curro FA. Clinical evaluation of ferric oxalate in relieving dentine hypersensitivity. J Oral Rehabil. 2004 Mar;31(3):245-50. doi: 10.1046/j.0305-182X.2003.01230.x. PMID 15025657
- [Background] Ide M, Morel AD, Wilson RF, Ashley FP. The role of a dentine-bonding agent in reducing cervical dentine sensitivity. J Clin Periodontol. 1998 Apr;25(4):286-90. doi: 10.1111/j.1600-051x.1998.tb02442.x. PMID 9565278
- [Background] Kakaboura A, Rahiotis C, Thomaidis S, Doukoudakis S. Clinical effectiveness of two agents on the treatment of tooth cervical hypersensitivity. Am J Dent. 2005 Aug;18(4):291-5. PMID 16296439
- [Background] Kerns DG, Scheidt MJ, Pashley DH, Horner JA, Strong SL, Van Dyke TE. Dentinal tubule occlusion and root hypersensitivity. J Periodontol. 1991 Jul;62(7):421-8. doi: 10.1902/jop.1991.62.7.421. PMID 1920008
- [Background] Levitch LC, Bader JD, Shugars DA, Heymann HO. Non-carious cervical lesions. J Dent. 1994 Aug;22(4):195-207. doi: 10.1016/0300-5712(94)90107-4. PMID 7962894
- [Background] LittleStar ML, Summitt JB. Non-carious cervical lesions: an evidenced-based approach to their diagnosis. Tex Dent J. 2003 Oct;120(10):972-80. No abstract available. PMID 14619725
- [Background] Lussi A, Schaffner M. Progression of and risk factors for dental erosion and wedge-shaped defects over a 6-year period. Caries Res. 2000 Mar-Apr;34(2):182-7. doi: 10.1159/000016587. PMID 10773637
- [Background] Lyttle HA, Sidhu N, Smyth B. A study of the classification and treatment of noncarious cervical lesions by general practitioners. J Prosthet Dent. 1998 Mar;79(3):342-6. doi: 10.1016/s0022-3913(98)70248-3. PMID 9553890
- [Background] Miller E, Deleger S, Murphy J (2002). Implementing and managing adaptive designs for clinical trials. http://www.pharmaceutical-int.com/categories/interactive-clinical-technologies-inc/implementing-and-managing-adaptive-designs-for-clinical-trials.asp.
- [Background] American Academy of Operative Dentistry. Non-carious cervical lesions. Recommendations for clinical practice. Oper Dent. 2003 Mar-Apr;28(2):109-13. No abstract available. PMID 12670064
- [Background] Ommerborn MA, Schneider C, Giraki M, Schafer R, Singh P, Franz M, Raab WH. In vivo evaluation of noncarious cervical lesions in sleep bruxism subjects. J Prosthet Dent. 2007 Aug;98(2):150-8. doi: 10.1016/S0022-3913(07)60048-1. PMID 17692596
- [Background] Osborne-Smith KL, Burke FJ, Wilson NH. The aetiology of the non-carious cervical lesion. Int Dent J. 1999 Jun;49(3):139-43. doi: 10.1002/j.1875-595x.1999.tb00898.x. PMID 10858746
- [Background] Pamir T, Dalgar H, Onal B. Clinical evaluation of three desensitizing agents in relieving dentin hypersensitivity. Oper Dent. 2007 Nov-Dec;32(6):544-8. doi: 10.2341/07-5. PMID 18051003
- [Background] Prati C, Cervellati F, Sanasi V, Montebugnoli L. Treatment of cervical dentin hypersensitivity with resin adhesives: 4-week evaluation. Am J Dent. 2001 Dec;14(6):378-82. PMID 11949798
- [Background] Rees JS. The biomechanics of abfraction. Proc Inst Mech Eng H. 2006 Jan;220(1):69-80. doi: 10.1243/095441105X69141. PMID 16459447
- [Background] Rimondini L, Baroni C, Carrassi A. Ultrastructure of hypersensitive and non-sensitive dentine. A study on replica models. J Clin Periodontol. 1995 Dec;22(12):899-902. doi: 10.1111/j.1600-051x.1995.tb01792.x. PMID 8613556
- [Background] Tavss EA, Fisher SW, Campbell S, Bonta Y, Darcy-Siegel J, Blackwell BL, Volpe AR, Miller SE. The scientific rationale and development of an optimized dentifrice for the treatment of dentin hypersensitivity. Am J Dent. 2004 Feb;17(1):61-70. PMID 15241912
- [Background] Telles D, Pegoraro LF, Pereira JC. Prevalence of noncarious cervical lesions and their relation to occlusal aspects: a clinical study. J Esthet Dent. 2000;12(1):10-5. doi: 10.1111/j.1708-8240.2000.tb00193.x. PMID 11323828
- [Background] Trowbridge HO, Silver DR. A review of current approaches to in-office management of tooth hypersensitivity. Dent Clin North Am. 1990 Jul;34(3):561-81. PMID 2197128
- [Background] Tyas MJ. The Class V lesion--aetiology and restoration. Aust Dent J. 1995 Jun;40(3):167-70. doi: 10.1111/j.1834-7819.1995.tb05631.x. PMID 7661762
- [Background] Yates RJ, Newcombe RG, Addy M. Dentine hypersensitivity: a randomised, double-blind placebo-controlled study of the efficacy of a fluoride-sensitive teeth mouthrinse. J Clin Periodontol. 2004 Oct;31(10):885-9. doi: 10.1111/j.1600-051X.2004.00581.x. PMID 15367193
- [Background] Zantner C, Popescu O, Martus P, Kielbassa AM. Randomized clinical study on the efficacy of a new lacquer for dentine hypersensitivity. Schweiz Monatsschr Zahnmed. 2006;116(12):1232-7. PMID 17233322
- [Background] Johansson A, Haraldson T, Omar R, Kiliaridis S, Carlsson GE. A system for assessing the severity and progression of occlusal tooth wear. J Oral Rehabil. 1993 Mar;20(2):125-31. doi: 10.1111/j.1365-2842.1993.tb01596.x. PMID 8468624
- [Background] Lavigne GJ, Manzini C, Kato T (2005). Sleep Bruxism. In: Principles and practice of sleep medicine. MH Kryger, T Roth and WC Dement editors. Philadelphia: Elsevier, pp. 946-59
- [Derived] Curro FA, Vena D, Naftolin F, Terracio L, Thompson VP. The PBRN initiative: transforming new technologies to improve patient care. J Dent Res. 2012 Jul;91(7 Suppl):12S-20S. doi: 10.1177/0022034512447948. PMID 22699662